CLINICAL TRIAL: NCT03584269
Title: Non Invasive Ventilation and Nocturnal Alveolar Hypoventilation in Patients With Chronic Obstructive Pulmonary Disease (COPD) Treated by Long Term Oxygen Therapy at Home
Brief Title: Innovation in NOn Invasive Ventilation in COPD Patients Treated by Long Term Oxygen Therapy
Acronym: INOV-LTOT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruiting difficulties
Sponsor: University Hospital, Grenoble (Other)
Collaborators: AGIR à Dom (Other); ResMed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 38RC17.117
Record Dates: First submitted 2018-01-22; First posted 2018-07-12 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Oxygenation Long term; Non invasive Ventilation; Nocturnal Hypoventilation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NIV Device + LTOT (Experimental): administration of ventilary support, without using an invasive artificial airway
  Interventions: Device: NIV Device + LTOT
- LTOT (Active Comparator): standard treatment, without NIV
  Interventions: Device: LTOT

INTERVENTIONS:
Device: NIV Device + LTOT — Respiratory assistance by a facial mask without intubation or tracheotomy
  Arms: NIV Device + LTOT
Device: LTOT — Long term oxygenatory tyherapy without NIV
  Arms: LTOT

SUMMARY:
The aim of this study is to investigate the efficacy of non-invasive ventilation (NIV) on nocturnal hypoventilation in patients with chronic obstructive pulmonary disease (COPD) who are on long term oxygen therapy (LTOT) at home.

DETAILED DESCRIPTION:
This is a prospective, randomized, open labelled study. The primary outcome is nocturnal transcutaneous CO2 (PtCO2) after 3 months of non-invasive ventilation. Three hundred COPD patients on LTOT will be screened and assessed by pulmonary function tests, blood gases and nocturnal PtCO2 at their home. This will allow the determination of the prevalence of nocturnal hypoventilation in COPD patients on LTOT (a secondary outcome) and to select patients who meet the inclusion criteria for the RCT and randomization to NIV + LTOT or to continue LTOT alone (n=38). Patients will undergo the same assessments at the end of the three-month intervention period.

ELIGIBILITY:
Inclusion Criteria:

* chronic obstructive pulmonary disease (COPD)

  * on long term oxygen therapy (LTOT)
  * affiliated to French social security system or equivalent
  * informed consent signed

Exclusion Criteria:

* Diurnal PtCO2 >55mmHg
* Patient who has had an exacerbation of COPD requiring a change in management or treatment in the last 4 weeks prior to the inclusion visit.
* Pregnant or breathfeeding women
* Prisonners or persons who require protection by the law
* Exclusion period from another study
* Persons who, according to the investigator, are expected no to meet all study obligations

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-06-28 (Actual); Primary Completion 2018-07-09 (Actual); Study Completion 2019-09-23 (Actual)

PRIMARY OUTCOMES:
Nocturnal transcutaneous pressure CO2 (PtCO2) | 3 months
  Measurement of nocturnal PtCO2 using the SenTec system

SECONDARY OUTCOMES:
Saint George's Respiratory Questionnaire | 3 months
  Measure of quality of life
FEV1 | 3 months
  Pulmonary function tests
Vital capacity | 3 months
  Pulmonary function tests
PaO2 | 3 months
  Blood gases
PaCO2 | 3 months
  Blood gases
Steps per day | 3 months
  Physical activity measured at home (one week)
Time in supine and sitting positions | 3 months
  Physical activity measured at home (one week)
Energy expenditure | 3 months
  Physical activity measured at home (one week)
Heart Rate | 3 months
  Physiological responses during the Semi paced 3-min Chair rise test
SaO2 | 3 months
  Physiological responses during the Semi paced 3-min Chair rise test
Dyspnea score | 3 months
  Symptoms during the Semi paced 3-min Chair rise test
Fatigue score | 3 months
  Symptoms during the Semi paced 3-min Chair rise test
Cholesterol | 3 months
  Biological parameters
Triglycerides | 3 months
  Biological parameters
Fasting Glucose | 3 months
  Biological parameters
CRPus | 3 months
  Biological parameters
HBA1c | 3 months
  Biological parameters

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis Pépin, Pr, PhD, Principal Investigator — University Grenoble Hospital
Locations (1):
- University Hospital Grenoble, La Tronche, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ko FW, Chan KP, Hui DS, Goddard JR, Shaw JG, Reid DW, Yang IA. Acute exacerbation of COPD. Respirology. 2016 Oct;21(7):1152-65. doi: 10.1111/resp.12780. Epub 2016 Mar 30. PMID 27028990
- [Result] Dretzke J, Moore D, Dave C, Mukherjee R, Price MJ, Bayliss S, Wu X, Jordan RE, Turner AM. The effect of domiciliary noninvasive ventilation on clinical outcomes in stable and recently hospitalized patients with COPD: a systematic review and meta-analysis. Int J Chron Obstruct Pulmon Dis. 2016 Sep 16;11:2269-2286. doi: 10.2147/COPD.S104238. eCollection 2016. PMID 27698560
- [Result] Borel JC, Pepin JL, Pison C, Vesin A, Gonzalez-Bermejo J, Court-Fortune I, Timsit JF. Long-term adherence with non-invasive ventilation improves prognosis in obese COPD patients. Respirology. 2014 Aug;19(6):857-65. doi: 10.1111/resp.12327. Epub 2014 Jun 9. PMID 24912564
- [Result] Kohnlein T, Windisch W, Kohler D, Drabik A, Geiseler J, Hartl S, Karg O, Laier-Groeneveld G, Nava S, Schonhofer B, Schucher B, Wegscheider K, Criee CP, Welte T. Non-invasive positive pressure ventilation for the treatment of severe stable chronic obstructive pulmonary disease: a prospective, multicentre, randomised, controlled clinical trial. Lancet Respir Med. 2014 Sep;2(9):698-705. doi: 10.1016/S2213-2600(14)70153-5. Epub 2014 Jul 24. PMID 25066329
- [Result] Meecham Jones DJ, Paul EA, Jones PW, Wedzicha JA. Nasal pressure support ventilation plus oxygen compared with oxygen therapy alone in hypercapnic COPD. Am J Respir Crit Care Med. 1995 Aug;152(2):538-44. doi: 10.1164/ajrccm.152.2.7633704.